CLINICAL TRIAL: NCT00805701
Title: Randomized, Double-Blind, Placebo-Controlled Trial Assessing The Efficacy And Safety Of Dutasteride At Improving Lower Urinary Tract Symptoms In Men With Clinically Localized Prostate Cancer Being Treated With Single-Dose Goserelin, Trans-Urethral Incision Of Prostate, And Interval Brachytherapy
Brief Title: Study Assessing The Efficacy And Safety Of Avodart (Dutasteride) At Improving Urinary Symptoms In Men With Prostate Cancer Who Are Undergoing Seed Implantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bay State Clinical Trials, Inc. (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: 047838
Record Dates: First submitted 2008-12-05; First posted 2008-12-10 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; avodart; dutasteride; mitcheson
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 0.5mg Avodart (Active Comparator): .5mg avodart capsule orally once a day during 13 months
  Interventions: Drug: avodart
- Placebo (Placebo Comparator): placebo capsule orally daily for 13 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: avodart — 0.5 avodart once daily for 13 weeks
  Other Names: dutasteride
  Arms: 0.5mg Avodart
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
Avodart (dutasteride) reduces the male hormone (DHT) that leads to prostate growth and stimulates cancerous growth. Avodart is currently approved by the FDA to treat men with symptoms of an enlarged prostate. Avodart works by reducing DHT and prostate size; therefore, the drug may be useful in improving lower urinary tract symptoms (LUTS) such as frequency, urgency, weak stream, and urination difficulty (dysuria), among others, in men with prostate cancer. Avodart may be effective in men with prostate cancer who are being treated with hormonal therapy with one injection of Zolodex (goserelin) followed one month later with a trans-urethral incision of the prostate (TUIP), and three months after that, seed implantation (SI) of the prostate.

The purpose of this study is to test whether Avodart (dutasteride) is effective on LUTS and dysuria in men with localized prostate cancer being treated with single-dose goserelin, TUIP, and interval SI.

DETAILED DESCRIPTION:
Dutasteride is an inhibitor of the 5 alpha reductase type I and type II enzymes that convert testosterone to DHT, the male hormone that leads to benign prostate growth and drives malignant growth. Dutasteride has been shown to significantly decrease intraprostatic DHT in men with localized prostate cancer, and additionally cause apoptosis and regression of some prostate cancers [Andriole, 2004a; Andriole, 2004b]. Furthermore, reduction in tumor volume has also been demonstrated in human prostate tissue [Iczkowski, 2004]. Dutasteride is currently indicated to treat symptomatic BPH in men with enlarged prostates, but is also being studied to reduce the risk of prostate cancer in men at risk (elevated PSA and previous negative biopsy). Dutasteride is clinically useful at improving lower urinary tract symptoms (LUTS) in men with clinically-localized prostate cancer and voiding difficulty being treated with single-dose goserelin, TUIP, and interval SI. [Mitcheson, personal observation].

ELIGIBILITY:
Inclusion Criteria:A subject will be eligible for inclusion in this study only if all of the following criteria apply:

1. Must be male ≥35 and ≤90 years of age
2. Have biopsy proven, localized prostate cancer
3. Gleason score ≤ 8
4. Clinical stage T1c-T2b
5. Serum PSA (prostate specific antigen) ≤10ng/mL within the 12 months period prior to positive prostate biopsy.
6. Able to swallow and retain oral medication
7. Able and willing to participate in the full duration of the study
8. Able to read and write (health outcomes questionnaires are self-administered), understand instructions related to study procedures and give written informed consent.

Exclusion Criteria:

1. Subject has ever been treated for prostate cancer with any of the following:

   * Radiotherapy (external beam or brachytherapy)
   * Chemotherapy
   * Hormonal therapy (e.g., megestrol, medroxyprogesterone, cyproterone, diethyl-stilbestrol (DES)
   * Oral glucocorticoids
   * Gonadotropin Releasing Hormone (GnRH) analogues (e.g., leuprolide, goserelin) other than the single-dose gosereline given as treatment in this study.
2. Glucocorticoids, except inhaled or topical, are not permitted within 3 months prior to visit one
3. Current and/or previous use of the following medications:

   * Finasteride (Proscar, Propecia), or Dutasteride (Avodart) exposure within 6 months prior to study entry are excluded.
   * Any other investigational 5-reductase inhibitors within the past 12 months.
   * Anabolic steroids (subject must discontinued for 6 months prior to study entry to be eligible)
   * Drugs with antiandrogenic properties within the past 6 months (e.g,. spironolactone, flutamide, bicalutamide, *cimetidine, *ketoconazole, progestational agents) *The use of cimetidine is permitted prior to study entry. The use of topical ketoconazole is permitted prior to and during the study.

Ages: 35 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the effect of dutasteride on dysuria, voiding and LUTS | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: Henry D Mitcheson, MD, Principal Investigator — Bay State Clinical Trials, Inc.
Locations (1):
- Bay State Clinical Trials, Inc., Watertown, Massachusetts, United States